CLINICAL TRIAL: NCT02866656
Title: The Clinical Research of Low Intensity Continuous Ultrasonic on Lower Limb Arteriosclerosis Occlusion(ASO) Syndrome
Brief Title: The Clinical Research of Low Intensity Continuous Ultrasonic on Lower Limb Arteriosclerosis Occlusion（ASO） Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Junli Duan, Deputy director of the department of Gerontology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-16-007
Record Dates: First submitted 2016-04-12; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Arteriosclerosis
MeSH Terms: conditions — Arteriosclerosis | interventions — Ultrasonic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Experimental): patients were given Conventional conservative treatment；
  Interventions: Other: Conventional conservative treatment
- therapeutic ultrasound group (Experimental): patients were given Conventional conservative treatment and low intensity ultrasonic treatment ；
  Interventions: Other: Conventional conservative treatment; Device: therapeutic ultrasound

INTERVENTIONS:
Other: Conventional conservative treatment — Treatment last for 4 weeks, three times a week,
Device: therapeutic ultrasound — Treatment last for 4 weeks, three times a week, stimulation was given 8 minutes every time, location of treatment were lower limb ischemia area and its surrounding tissues；
  Arms: therapeutic ultrasound group

SUMMARY:
In the present study, by evaluating the efficacy and safety of low intensity ultrasonic on ASO, to explore the noninvasive auxiliary treatment of ASO. 90 patients were randomly divided into 2 groups: A)control group, patients were given Conventional conservative treatment; B）treatment group, patients were given Conventional conservative treatment and low intensity ultrasonic treatment ; Treatments last for 4 weeks, three times a week, stimulation was given 8 minutes every time, location of treatment were lower limb ischemia area and its surrounding tissues; outcome indicators were recorded Before and 4 weeks after the trial, The Walking Impairment Questionnaire (WIQ), ankle brachial ratio, the farthest distance Walking, percutaneous tissue oxygen tension, tissue oxygenation index recovery time, local skin temperature, ultrasonic blood vessels, and muscle enzymes, hepatic and kidney function.

DETAILED DESCRIPTION:
Ultrasound is a form of sound whose frequency is higher than the natural audible range for humans (> 20 kHz) and ultrasonography has been widely used as diagnostic devices for several decades. In addition to diagnostic purposes, ultrasound is clinically used for therapeutic applications, including tumor ablation, thrombolysis, bone regeneration, and facilitated drug delivery. Recently, therapeutic angiogenic effects of low-intensity ultrasound have been reported in endothelial cells, chick chorioallantoic membrane, and a rat model of hind limb ischemia. the investigators hypothesis low-intensity ultrasound can improve the ailment of ASO. In the present study, by evaluating the efficacy and safety of low intensity ultrasonic on ASO, to explore the noninvasive auxiliary treatment of ASO. 90 patients were randomly divided into 2 groups: A)control group，patients were given Conventional conservative treatment: B）treatment group，patients were given Conventional conservative treatment and low intensity ultrasonic treatment; Treatments last for 4 weeks, three times a week, stimulation was given 8 minutes every time, location of treatment were lower limb ischemia area and its surrounding tissues；outcome indicators were recorded Before and 4 weeks after the trial, The Walking Impairment Questionnaire (WIQ), ankle brachial ratio, the farthest distance Walking, percutaneous tissue oxygen tension, tissue oxygenation index recovery time, local skin temperature, ultrasonic blood vessels, and muscle enzymes, hepatic and kidney function.

the investigators speculate after 4 weeks of Low intensity ultrasonic treatment, all the observation index of ASO patients can be improved; meanwhile, creatine kinase, liver and kidney function, blood in urine routine, electrocardiogram (ecg) has no obvious change.

ELIGIBILITY:
Inclusion Criteria:

* lower limb arteriosclerosis occlusion disorder patients
* In line with the Fontaine II - Ⅲ period clinical stage
* Aged 35 to 70 years old
* No major organ dysfunction, including heart, liver and kidney
* Can understand the procedures and methods of the test, strictly observe clinical trial plan to complete the test, and sign the informed consent

Exclusion Criteria:

* Fontaine clinical staging in patients with stage I
* Aged under 35 or more than 70 - year - old patient
* Women with pregnancy or lactation
* Childless and one year plan pregnancy
* Patients with cardiac pacemaker
* Patients with malignant tumor, psychosis
* Accompanied by severe heart, brain, kidney and hematopoietic system disease
* The following appeared in the process of being test: myocardial infarction, severe/unstable angina, coronary artery/peripheral artery bypass grafts, heart failure, cerebrovascular accident (including transient ischemic attack); And epilepsy, severe liver and kidney function is not complete, mechanical intestinal obstruction, bradycardia, bronchial asthma and other diseases
* Researchers think the patient has any problem that may cause the participants can't finish this research ，or any other situation of risk to participants

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Improvement of ankle brachial ratio at 4 weeks of treatment | 4weeks

SECONDARY OUTCOMES:
Improvement of local skin temperature at 4 weeks of treatment | 4weeks
Recovery of ultrasonic blood vessels at 4 weeks of treatment | 4weeks
Enhancement of the value of muscle enzymes at 4 weeks of treatment | 4weeks
Elevation of the value of hepatic and kidney function at 4 weeks of treatment | 4weeks
Improvement of the farthest distance Walking at 4 weeks of treatment | 4weeks
Changes of percutaneous tissue oxygen tension at 4 weeks of treatment | 4weeks

IPD SHARING:
Plan to Share IPD: Undecided